CLINICAL TRIAL: NCT05796349
Title: Study on Data Acquisition and Image Characteristics of Brain Multifrequency EIT in Healthy People and Patients With Brain Diseases
Status: Completed | Type: Observational
Sponsor: Jieshi Ma (Other Government)
Responsible Party: Sponsor-Investigator, Jieshi Ma, Deputy Director of MedicaEngineering Department, Army Medical Center of PLA
Organization: Army Medical Center of PLA (Other Government)
Other Study IDs: AMCPLA
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Cerebral Hemorrhage; Cerebral Ischemia; Cerebral Edema; Healthy
Keywords: Multifrequency electrical impedance tomography; Intracranial abnormality; Detection; Symmetry
MeSH Terms: conditions — Cerebral Hemorrhage; Brain Ischemia; Brain Edema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy group: The healthy group included 16 individuals (male, age 40.25±11.18). No history of brain disease and no abnormalities were seen on plain CT scans of their brains.
  Interventions: Diagnostic Test: multifrequency EIT-based for detecting intracranial abnormalities
- patient group: The patient group included 8 patients with brain diseases (7 males, age 59±10.46). Obvious lesions were visible on the patients' CT or MRI images, including 6 patients with intracranial hemorrhage, 1 patient with cerebral ischemia, and 1 patient with cerebral edema
  Interventions: Diagnostic Test: multifrequency EIT-based for detecting intracranial abnormalities

INTERVENTIONS:
Diagnostic Test: multifrequency EIT-based for detecting intracranial abnormalities — For subjects who received clinical trials, 16 electrodes were placed equidistantly in their head, and brain EIT data were measured at 9 frequencies in the range of 21 kHz to 100 kHz by applying a current RMS of 176 microamps.MFEIT image sequences were obtained according to certain imaging algorithms.

SUMMARY:
The goal of this observational study is to compare the differences in the features of cerebral multifrequency EIT(cMFEIT) images between healthy subjects and patients with brain diseases and to explore the possibility of applying multifrequency EIT to intracranial abnormality detection.16 healthy volunteers and 8 patients with brain diseases were recruited as experimental subjects, and the cerebral EIT data of 9 frequencies in the range of 21 kHz - 100 kHz of all subjects were acquired with an EH-300 MFEIT system.

DETAILED DESCRIPTION:
For subjects who received clinical trials, 16 electrodes were placed equidistantly in their head, and brain EIT data were measured at 9 frequencies in the range of 21 kHz to 100 kHz by applying a current RMS of 176 microamps. The healthy group included 16 individuals (male, age 40.25±11.18). No history of brain disease and no abnormalities were seen on plain CT scans of their brains. Cerebral EIT data collection from healthy volunteers was performed in a dedicated laboratory with temperature controlled at 24±1 °C and 52%±1% humidity in 2022. The subjects were lying in a horizontal position. The patient group included 8 patients with brain diseases (7 males, age 59±10.46). Obvious lesions were visible on the patients' CT or MRI images, including 6 patients with intracranial hemorrhage, 1 patient with cerebral ischemia, and 1 patient with cerebral edema. Data from patients with brain diseases were collected at the neurosurgical intensive care unit at the Army Medical Center of PLA in 2022. The cerebral EIT data of the patients were collected in the same position as the healthy individuals. The MFEIT image sequence is obtained according to a certain imaging algorithm, and the ROI area ratio (AR_ROI) on the left and right sides of the image and the average value of the reconstructed ROI resistivity change (MVRRC_ROI) are extracted. Based on the extracted indicators, the geometric asymmetry index (GAI) and intensity asymmetry index (IAI) was further proposed to characterize the symmetry of MFEIT images, and the differences between the two groups of subjects on MFEIT images were statistically compared and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Health Group: No history of brain disease and no abnormalities were seen on plain CT scans of their brains.
2. Patient Group: Patients with cerebral hemorrhage, cerebral ischemia, and cerebral edema, less than 12 days after onset.

Exclusion Criteria:

1. Health Group:

   * Neurological diseases such as epilepsy, brain tumors, and cerebral vascular malformations;
   * Neurological symptoms such as headache and dizziness;
   * Abnormal signals detected on CT.
2. Patient Group:

   * With other brain diseases without cerebral hemorrhage, cerebral ischemia, or brain edema;
   * With open craniocerebral injury;
   * With severe agitation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Health Group: No history of brain disease and no abnormalities were seen on plain CT scans of their brains.
  Patient Group: Obvious lesions were visible on the patient's CT or MRI images.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Whether there is a significant difference in the characteristic indicators (such as symmetry indicators) of multifrequency EIT images between healthy individuals and patients with brain diseases. | Up to 12 days after the patient's onset
  When there are significant differences in these indicators (such as symmetry indicators) (p<0.05), there is no need for further data collection

CONTACTS AND LOCATIONS:
Locations (1):
- PLA Army Characteristic Medical Center, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code